CLINICAL TRIAL: NCT05339386
Title: Developing Hyperpolarized 129Xe MRI Biomarkers for Evaluation of Pulmonary Arterial Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: 00148587
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (10 mL) will be collected from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiating Therapy: PAH patients who are newly initiating background therapy to treat pulmonary arterial hypertension.
  Interventions: Drug: Hyperpolarized Xe129
- Stable: PAH patients who are stable on therapy (On stable doses of background PAH therapy and diuretics for at least 90 days prior to screening).
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Lung MRI using gaseous contrast agent hyperpolarized 129Xe.
  Other Names: Xenon MRI; HP Xenon; 129Xe

SUMMARY:
In this study, hyperpolarized 129Xe MRI will be used to evaluate treatment efficacy in patients with pulmonary arterial hypertension (PAH). Participants will be imaged at 4 timepoints (baseline, 6 weeks post-therapy initiation, 12 weeks, and 18 weeks). Images will be analyzed to develop new biomarkers and to understand treatment effects.

DETAILED DESCRIPTION:
1. Optimize Xe-MRI Oscillation Imaging for PAH. Regional mapping of oscillations in the xenon RBC signal is a new technique that may provide new insights into microvascular function in PH. Recent innovations in Xe-MRI have enabled improvements to this methodology, but these have yet to be explored and optimized.
2. Quantify the short- and long-term repeatability of Xe-MRI oscillation imaging in patients with PAH. Hyperpolarized 129Xe oscillation imaging is a novel technique that may provide regional quantification of pulmonary microvascular function. However, the repeatability of this technique has not been measured, which limits its use as an outcome measure.
3. Determine the minimum time-point at which Xe-MRI shows a clinically meaningful change following treatment. Current standards in the PAH community are to assess treatment efficacy in PAH patients at 3-6 months using 6MWTs, REVEAL Lite scores, echocardiograms, and possibly RHCs. However, Xe-MRI may be more sensitive to functional improvements. We hypothesize that Xe-MRI biomarkers will show a clinically meaningful change within 12 weeks of initiation of pulmonary vasodilators.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming the diagnosis of WHO PAH Group 1 in any of the following subtypes:

  * Idiopathic PAH
  * Heritable PAH
  * Drug/toxin-induced PAH
  * PAH associated with CTD
* Symptomatic PAH classified as WHO FC I, II, or III.
* Documented Historical RHC with a mPAP ≥ 20 mmHg, PCWP ≤15 mmHg, and PVR ≥ 3 Wood Units (WU)
* Ability to adhere to the study visit schedule, adhere, and comply with all protocol requirements.
* Ability to understand and provide written informed consent.

For patients in the Initiating Therapy Arm:

* Initiation of pulmonary vasodilator therapy within ±3 weeks of baseline imaging timepoint.

For patients in the Stable Arm:

* On stable doses of background PAH therapy and diuretics (i.e., patient-specific dose goal for each therapy already achieved) for at least 90 days prior to screening; for infusion prostacyclins, dose adjustment within 10% of optimal dose is allowed per medical practice

Exclusion Criteria:

* Subject unable to undergo MRI based on MRI safety screening
* Diagnosis of pulmonary hypertension WHO Groups 2, 3, 4, or 5
* Pregnant or breastfeeding female subjects
* Prisoners or incarcerated individuals
* Any major surgical procedure within 90 days prior to study enrollment or planned surgical procedure during the study period.
* Concomitant medical disorder, condition, or history, that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent or would confound the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants to be enrolled will include individuals with diagnosed pulmonary arterial hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in RBC/Membrane Ratio | 18 weeks
  Absolute change over 4 imaging timepoints of RBC/Membrane Ratio from xenon MRI.

SECONDARY OUTCOMES:
Change in Xenon RBC uptake | 18 weeks
  Absolute change over 4 imaging timepoints of RBC/Gas ratio from xenon MRI.
Change in Xenon RBC oscillation amplitude | 18 weeks
  Absolute change over 4 imaging timepoints of RBC oscillation amplitude from xenon MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Niedbalski, PHD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request, deidentified subject data, including xenon MRI images may be shared with other researchers.